CLINICAL TRIAL: NCT04251156
Title: Effect and Safety of Semaglutide 2.4 mg Once-weekly on Weight Management in Subjects With Overweight or Obesity.
Brief Title: Research Study of How Well Semaglutide Works in People Living With Overweight or Obesity.
Acronym: STEP7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4379; U1111-1212-2189 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental): Once-weekly injections of gradually increased doses of semaglutide
  Interventions: Drug: Semaglutide
- Placebo (semaglutide) (Placebo Comparator): Once-weekly injections of gradually increased doses of semaglutide placebo
  Interventions: Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide administered subcutaneously (s.c., under the skin) as well as diet and physical activity counselling for 44 weeks. Doses gradually increased to 2.4 mg
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Semaglutide placebo administered s.c. as an adjunct to a reduced-calorie diet and increased physical activity regimen for 44 weeks
  Arms: Placebo (semaglutide)

SUMMARY:
This study will look at the change in body weight from the start to the end of the study. The purpose of the study is to compare the effect on body weight in people taking semaglutide (a new medicine) and people taking "dummy" medicine. In addition to taking the medicine participants will have talks with study staff about healthy food choices, how to be more physically active and what else they can do to lose weight. Participants will either get semaglutide or "dummy medicine" - which treatment is decided by chance. Participants will need to take 1 injection once a week. The study medicine is injected with a thin needle in a skinfold in the stomach, thigh or upper arm.• The study will last for about 1 year. Participants will have 11 clinic visits and 8 phone calls with the study doctor. Participants will have 3 clinic visits where they cannot eat and drink (water is allowed) for up to 8 hours before the visit and 1 clinic visit where they cannot eat and drink for up to 2 hours before the visit. (4 visits and 1 visit, respectively, if they have type 2 diabetes (T2D)). Participants will have 4 clinic visits where they will have blood samples taken. (5 visits if they have T2D). For China: Participants will have 9 clinic visits where they will have blood samples taken. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at the time of signing informed consent
* History of at least one self-reported unsuccessful dietary effort to lose body weight

For subjects without T2D at screening:

* Body mass index (BMI) of :
* greater than or equal to 30 kg/m^2
* greater than or equal to 27 kg/m^2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease

For subjects with T2D at screening:

* Diagnosed with T2D above or equal to 180 days prior to the day of screening
* Treated with either:
* diet and exercise alone or
* stable treatment (same drug(s), dose and dosing frequency) for at least 60 days prior to the day of screening with up to 3 oral antidiabetic medications alone or in any combination (metformin, α-glucosidase inhibitor (AGI), SU, glinides, SGLT2i or glitazone) according to local label
* HbA1c 7.0-10.0% (53-86 mmol/mol) (both inclusive)
* BMI greater than or equal to 27 kg/m^2

Exclusion Criteria:

* A self-reported change in body weight above 5 kg (11 lbs) within 90 days before screening irrespective of medical records

For subjects without T2D at screening:

- HbA1c equal to or above 6.5% (48 mmol/mol) as measured by the central laboratory at screening

For subjects with T2D at screening :

* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of below 30 mL/min/1.73 m^2 (below 60 mL/min/1.73 m^2 in subjects treated with SGLT2i) according to CKDEPI creatinine equation as defined by KDIGO 2012 by the central laboratory at screening
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor & Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (33):
- Brazil (2):
  - Instituto de Ciências Farmacêuticas de Estudos e Pesquisas, Aparecida de Goiânia, Goiás
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
- China (28):
  - The First Affiliated Hospital of Anhui Medical University-Endocrinology, Hefei, Anhui
  - Chinese People's Liberation Army General Hospital-Endocrinology, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital-Endocrinology, Fuzhou, Fujian
  - Cangzhou People's Hospital-Endocrinology, Cangzhou, Hebei
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - Harrison International Peace Hospital-Endocrinology, Hengshui, Hebei
  - Hengshui People's Hospital (Harrison International Peace Hospital)-Endocrinology, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University-Endocrinology, Shijiazhuang, Hebei
  - Inner Mongolia People's Hospital-Endocrinology, Hohhot, Inner Mongolia
  - The affiliated Hospital of Inner Mongolia Medical University-Endocrinology, Hohhot, Inner Mongolia
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - Jiangsu Province Hospital-Endocrinology, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - The First Bethune hospital of Jilin University-Endocrinology, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Huashan Hospital Fudan University-Endocrinology, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital (Tenth People's of Tongji University)-Endocrinology, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - Tongren Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- South Korea (2):
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Mu Y, Bao X, Eliaschewitz FG, Hansen MR, Kim BT, Koroleva A, Ma RCW, Yang T, Zu N, Liu M; STEP 7 Study Group. Efficacy and safety of once weekly semaglutide 2.4 mg for weight management in a predominantly east Asian population with overweight or obesity (STEP 7): a double-blind, multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2024 Mar;12(3):184-195. doi: 10.1016/S2213-8587(23)00388-1. Epub 2024 Feb 5. PMID 38330988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 28 sites in 3 countries as follows (all sites screened and randomized): Region China (includes China mainland and Hong Kong) China mainland (23 sites) and Hong Kong (1 site), Brazil (2 sites) and South Korea (2 sites).
Pre-assignment Details: Participants were randomized in 2:1 ratio to receive 2.4 mg semaglutide subcutaneously (s.c.) or semaglutide matching placebo. The trial has a 44-week treatment period (16 weeks of dose escalation period and 28 weeks of maintenance period), followed by a 7-week follow-up period.
Groups:
- Semaglutide 2.4 mg: Participants initiated at a once weekly dose of 0.25 mg semaglutide s.c. followed a fixed-dose escalation regimen, with dose increasing every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), to reach maintenance dose after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg once-weekly for an additional 28 weeks until week 44 adjunct to a reduced calorie diet and increased physical activity.
- Placebo: Participants received placebo matched to semaglutide s.c. once weekly for 44 weeks
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Placebo
Started | 249 | 126
Full Analysis Set (FAS) | 249 | 126
Safety Analysis Set (SAS) | 249 | 126
Treated | 249 | 126
Completed | 244 | 121
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Placebo | Total
Number analyzed (Participants) | 249 | 126 | 375
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (11) | 40 (11) | 41 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 59 | 170
  Male | 138 | 67 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 11 | 37
  Not Hispanic or Latino | 223 | 115 | 338
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 225 | 115 | 340
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 22 | 9 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight (Percentage [%])
Description: Change from baseline at week 0 to week 44 in body weight (%) is presented.The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: Full Analysis Set (FAS) which comprised all randomized participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Percentage change | -12.5 (7.4) | -3.6 (5.9)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority — Responses were analysed using an analysis of covariance model with randomized treatment and type 2 diabetes status as factors and baseline body weight as covariate; p < 0.0001, ANCOVA; Treatment difference = -8.47, 95% CI 2-sided [-10.17 to -6.76]

2. Primary Outcome: Number of Participants Who Achieved Body Weight Reduction Greater Than or Equal (>=) to 5% (Yes/No)
Description: Number of participants who achieved >=5% weight reduction at week 44 for in-trial observation period is presented.In the reported data, 'Yes' infers the number of participants who have achieved greater than or equal to 5% weight reduction, whereas 'No' infers the number of participants who have not achieved greater than or equal to 5% weight reduction. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: FAS which comprised all randomized participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Participants
  Yes | 203 | 36
  No | 35 | 80
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Placebo; Treatment policy estimand; Test type: Superiority — Responses were analysed using a binary logistic regression model with randomized treatment and type 2 diabetes status as factors and baseline body weight as covariate; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 13.07, 95% CI 2-sided [7.40 to 23.10]

3. Secondary Outcome: Number of Participants Who Achieved Body Weight Reduction Greater Than or Equal (>=) to 10% (Yes/No)
Description: Number of participants who achieved >=10% weight reduction at week 44 for in-trial observation period is presented. In the reported data, 'Yes' infers the number of participants who have achieved greater than or equal to 10% weight reduction, whereas 'No' infers the number of participants who have not achieved greater than or equal to 10% weight reduction. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Participants
  Yes | 151 | 12
  No | 87 | 104

4. Secondary Outcome: Number of Participants Who Achieved Body Weight Reduction Greater Than or Equal (>=) to 15% (Yes/No)
Description: Number of participants who achieved >=15% weight reduction at week 44 for in-trial observation period is presented. In the reported data, 'Yes' infers the number of participants who have achieved greater than or equal to 15% weight reduction, whereas 'No' infers the number of participants who have not achieved greater than or equal to 15% weight reduction. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Participants
  Yes | 82 | 7
  No | 156 | 109

5. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Centimeter (cm) | -11.1 (7.2) | -3.8 (5.8)

6. Secondary Outcome: Change From Baseline in Body Weight (Kilogram [kg])
Description: Change in body weight from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Kilogram (kg) | -11.9 (7.3) | -3.4 (6.0)

7. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change in BMI from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Kilograms per square meter (kg/m^2) | -4.3 (2.6) | -1.2 (2.1)

8. Secondary Outcome: Number of Participants Who Achieved Body Weight Reduction Greater Than or Equal (>=) to 20% (Yes/No)
Description: Number of participants who achieved >=20% weight reduction at week 44 for in-trial observation period is presented. In the reported data, 'Yes' infers the number of participants who have achieved greater than or equal to 20% weight reduction, whereas 'No' infers the number of participants who have not achieved greater than or equal to 20% weight reduction. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Participants
  Yes | 34 | 2
  No | 204 | 114

9. Secondary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
Millimeters of mercury (mmHg) | -7 (12) | -2 (12)

10. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) - Physical Functioning Score
Description: SF-36 is a 36-item participants-reported survey of participants health that measures the partici-pants overall health-related quality of life (HRQoL). SF-36 questionnaire measured 8 domains of functional health and well-being as well as 2 component summary scores (physical component summary and mental component summary). This outcome measure shows results for 'physical functioning domain'. Physical function domain score ranges from 0 to 100, with higher values indicating better functional health and well-being. Change from baseline (week 0) in the domain scores were evaluated at week 44. These outcome measures were evaluated based on data from in-trial observation period which is the uninterrupted time interval from (week 0) to (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 237 | 116
Score on a scale | 1.3 (4.7) | 0.2 (5.7)

11. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life-Lite for Clinical Trials (IWQOL-Lite for CT) - Physical Function Domain (5-items) Score
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on participants quality of life within the context of clinical trials. IWQOL-Lite-CT is a 20-item questionnaire-based instrument used to assess the impact of body weight changes on participants overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite and physical function domain scores range from 0 to 100, with higher scores reflecting better levels of functioning. This outcome measure shows results for 'physical function domain'. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 115
Score on a scale | 8.0 (16.4) | 2.3 (18.5)

12. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) (Percentage [%])
Description: Change in glycosylated haemoglobin (HbA1c) (%) from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 235 | 111
Percentage of HbA1c | -0.8 (0.8) | -0.1 (0.8)

13. Secondary Outcome: Change From Baseline in HbA1c (Millimoles Per Mole [mmol/Mol])
Description: Change in HbA1c (mmol/mol) from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per mole (mmol/mol)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 235 | 111
Millimoles per mole (mmol/mol) | -8.9 (9.2) | -1.3 (8.3)

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) (Milligrams Per Deciliter [mg/dL])
Description: Change in fasting plasma glucose (mg/dL) from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 234 | 112
Milligrams per deciliter (mg/dL) | -18.9 (25.3) | -1.1 (18.7)

15. Secondary Outcome: Change From Baseline in FPG (Millimoles Per Liter [mmol/L])
Description: Change in FPG (mmol/L) from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 234 | 112
Millimoles per litre (mmol/L) | -1.1 (1.4) | -0.1 (1.0)

16. Secondary Outcome: Change From Baseline in Fasting Serum Insulin: Ratio to Baseline
Description: Change in fasting serum insulin measured as milli-international units per milliliter (mIU/mL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 235 | 110
Ratio of fasting serum insulin | 0.76 (57.3) | 0.98 (62.9)

17. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 238 | 116
mmHg | -4 (9) | -1 (9)

18. Secondary Outcome: Change From Baseline in Total Cholesterol: Ratio to Baseline
Description: Change in total cholesterol measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 112
Ratio of total cholesterol | 0.94 (17.5) | 1.04 (17.5)

19. Secondary Outcome: Change From Baseline in High-Density Lipoproteins (HDL)-Ratio to Baseline
Description: Change in HDL measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 111
Ratio of HDL | 1.05 (15.5) | 1.08 (16.6)

20. Secondary Outcome: Change From Baseline in Low-Density Lipoproteins (LDL)-Ratio to Baseline
Description: Change in LDL measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 110
Ratio of LDL | 0.97 (33.0) | 1.04 (29.0)

21. Secondary Outcome: Change From Baseline in Very Low-Density Lipoproteins (VLDL)-Ratio to Baseline
Description: Change in VLDL measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 111
Ratio of VLDL | 0.71 (45.3) | 0.96 (44.3)

22. Secondary Outcome: Change From Baseline in Free Fatty Acids-Ratio to Baseline
Description: Change in free fatty acids measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 110
Ratio of free fatty acids | 0.91 (66.9) | 1.05 (69.7)

23. Secondary Outcome: Change From Baseline in Triglycerides-Ratio to Baseline
Description: Change in triglycerides measured as milligrams per deciliter (mg/dL) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 112
Ratio of triglycerides | 0.71 (50.2) | 0.96 (52.6)

24. Secondary Outcome: Change From Baseline in SF-36 All Domains (Except Physical Functioning) and 2 Component Summary Scores
Description: SF-36 is a 36-item participant-reported survey of health that measures the overall HRQoL. SF-36 questionnaire measured 8 domains of functional health and well-being as well as 2 component summary scores (physical and mental component summary). This outcome measure shows results for all domains (except physical functioning) and 2 component summary scores. The score ranges from 0 to 100, with higher values indicating better functional health and well-being. Change from baseline week 0 in domain and component summary scores were evaluated at week 44 based on data from in-trial observation period which is uninterrupted time interval from (week 0) to (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 237 | 116
Score on a scale
  Role-Physical | 0.5 (5.1) | -0.8 (6.3)
  Bodily Pain | -0.3 (7.1) | -1.2 (7.3)
  General Health | 3.2 (7.6) | 1.6 (7.6)
  Vitality | 0.3 (7.8) | -1.1 (6.7)
  Social Functioning | -0.5 (5.6) | -0.5 (5.0)
  Role-Emotional | 0.5 (7.0) | -0.9 (5.9)
  Mental Health | -0.1 (7.4) | -1.8 (7.1)
  Physical component summary | 1.4 (5.2) | 0.4 (5.5)
  Mental component summary | -0.3 (7.1) | -1.5 (6.1)

25. Secondary Outcome: Change From Baseline in IWQOL-Lite for Physical Domain Score, Psychological Domain Score and Total Score
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on participants quality of life within the context of clinical trials. IWQOL-Lite-CT is a 20-item questionnaire-based instrument used to assess the impact of body weight changes on participants overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite scores for physical domain score, psychosocial domain score and total score ranges from 0 to 100, with higher scores reflecting better levels of functioning. This outcome measure shows results for 'physical and psychosocial domains, and for total'. The outcome measure was evaluated based on the data from in-trial observation period which is the uninterrupted time interval from start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 115
Score on a scale
  Physical | 7.2 (16.3) | 2.0 (18.3)
  Psychosocial | 12.0 (17.3) | 4.8 (17.4)
  Total | 10.3 (15.4) | 3.8 (16.2)

26. Secondary Outcome: Number of Participants Who Achieved Responder Definition Value for SF-36 Physical Functioning Score (Yes/No)
Description: The number of participants experiencing a meaningful within participant improvement in SF-36 Physical function after 44 weeks was determined based on 3.7 threshold. The threshold of 3.7 is specific for overweight or obese population included in the study and calculated using participant global rating anchor questionnaires to reflect participants own perspective based on Food and Drug Administration (FDA) recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers number of participants who have not achieved an improvement in score greater than or equal to the threshold. The outcome measure was evaluated based on in-trial observation period which is the uninterrupted time interval from start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 237 | 116
Participants
  Yes | 69 | 27
  No | 168 | 89

27. Secondary Outcome: Number of Participants Who Achieved Responder Definition Value For IWQoL-Lite for CT Physical Function (5-items) Score (Yes/No)
Description: The number of participants experiencing a meaningful within participant improvement in IWQOL-Lite-CT physical function after 44 weeks was determined based on thresholds of 14.6. The threshold of 14.6 is specific for the population with overweight or obesity included in the study and calculated using patient global rating anchor questionnaires to reflect participants own perspective based on FDA recommendations. In the reported data, "Yes" infers the number of participants who have achieved an improvement in score greater than or equal to the threshold and "No" infers the number of participants who have not achieved an improvement in score greater than or equal to the threshold. The outcome measure was evaluated based on in-trial observation period which is the uninterrupted time interval from start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 115
Participants
  Yes | 83 | 22
  No | 153 | 93

28. Secondary Outcome: Number of Participants With Type 2 Diabetes (T2D) Who Achieved HbA1c Less Than (<) 7.0 Percent (%) (53 mmol/Mol)
Description: Number of participants with T2D who achieved HbA1c < 7% (53 mmol/mol) at week 44 is presented. In the reported data, "Yes" infers the number of participants who have achieved HbA1c values less than the 7% and "No" infers the number of participants who have not achieved HbA1c values less than the 7%. The outcome measure was evaluated based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 62 | 28
Participants
  Yes | 57 | 8
  No | 5 | 20

29. Secondary Outcome: Number of Participants With T2D Who Achieved HbA1c Less Than or Equal to (<=) 6.5% (48 mmol/Mol)
Description: Number of participants with T2D who achieved HbA1c <= 6.5% (48 mmol/mol) at week 44 is presented. In the reported data, "Yes" infers the number of participants who have achieved HbA1c values less than or equal to 6.5% and "No" infers the number of participants who have not achieved HbA1c values less than or equal to 6.5%. The outcome measure was evaluated based on the data from in-trial observation period which was defined as the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: At week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 62 | 28
Participants
  Yes | 51 | 4
  No | 11 | 24

30. Secondary Outcome: Change From Baseline in Glycaemic Category (Normo-Glycaemia, Pre-Diabetes, T2D) in Participants With no T2D at Baseline
Description: Change from baseline in number of participants in glycaemic categories (normo-glycaemia, pre-diabetes and type 2 diabetes) at baseline (week 0) to week 44 are presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 173 | 84
Participants
  Normo-glycaemia | 158 | 53
  Pre-diabetes | 15 | 29
  Diabetes | 0 | 2

31. Secondary Outcome: Change From Baseline in Number of Participants With Antihypertensive Medication (Decrease, No Change, Increase)
Description: Change from baseline in number of participants in antihypertensive medication (decrease, no change, increase) at baseline (week 0) to week 44 are presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 242 | 118
Participants
  Decreased | 8 | 2
  No change | 57 | 23
  Increased | 9 | 4

32. Secondary Outcome: Change From Baseline in Number of Participants With Lipid-Lowering Medication (Decrease, No Change, Increase)
Description: Change from baseline in number of participants in lipid-lowering medication (decrease, no change, increase) at baseline (week 0) to week 44 are presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 242 | 118
Participants
  Decreased | 3 | 1
  No change | 31 | 13
  Increased | 1 | 4

33. Secondary Outcome: Change From Baseline in Number of Participants With Concomitant Oral Antidiabetic Medication (Decrease, No Change, Increase) in Participants With No T2D at Baseline
Description: Change from basline in number of participants with concomitant oral antidiabetic medication (decrease, no change, increase) at baseline (week 0) to week 44 are presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 63 | 30
Participants
  Decreased | 16 | 2
  No change | 35 | 16
  Increased | 1 | 6

34. Secondary Outcome: Change From Baseline in Number of Participants in Fatty Liver Index (FLI) Score Category
Description: Change from baseline in number of participants in fatty liver index (FLI) at baseline (week 0) to week 44 are presented. The fatty liver index is based on an algorithm including body mass index, waist circumference, triglycerides and gamma-glutamyl-transferase. The FLI scores less than (<) 30 indicates no hepatic steatosis (no fatty liver), FLI greater than or equal to (>=) 30 to less than (<) 60 indicates intermediate status of hepatic steatosis and >=60 indicates severe/worse hepatic steatosis. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 236 | 113
Participants
  <30 | 67 | 8
  30<= to <60 | 62 | 17
  >=60 | 107 | 88

35. Secondary Outcome: Number of Participants Who From Randomization Permanently Discontinued Randomized Trial Product
Description: Number of participants who permanently discontinued randomized trial product from baseline (week 0) to week 44 are presented. The outcome measure was evaluated based on the data from in-trial observation period. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to last trial-related participant-site contact (week 51).
Time Frame: Baseline (week 0), week 44
Population: FAS which comprised all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 249 | 126
Participants | 18 | 16

36. Secondary Outcome: Time to Permanent Discontinuation of Randomized Trial Product (Weeks)
Description: Time to permanent discontinuation of randomised trial product from baseline (week 0) to week 44 is reported. Participants who permanently discontinued the randomised trial product during the in-trial observation period were only included in the analysis. In-trial observation period: the uninterrupted time interval from the start of randomization (week 0) to date of last contact with trial site (week 51).
Time Frame: Baseline (week 0), week 44
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 18 | 16
Weeks | 16.7 [5.4 to 43.1] | 18.8 [3.0 to 43.3]

37. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned are treatment emergent adverse events (TEAE) defined as an event with onset during the on-treatment observation period. On-treatment observation period: the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0), week 51
Population: Safety Analysis Set (SAS) included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 249 | 126
Events | 1122 | 415

38. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. SAE results occurred from week 0 to week 51 is presented based on the on-treatment observation, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) plus a 7 week follow-up period and excluding any off-treatment time intervals. Off-treatment time interval: time period with at least two consecutive missed doses.
Time Frame: Baseline (week 0), week 51
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 249 | 126
Events | 14 | 8

39. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemia Episodes (Yes/No) in Participants With T2D at Week 0
Description: Hypoglycaemic episodes with onset during on-treatment observation period were considered treatment-emergent. Number of treatment emergent severe or BG confirmed symptomatic hypoglycaemia episodes in participants with T2D at week 0 with onset during on-treatment observation period were presented.
Time Frame: Baseline (week 0), week 51
Population: Analysis population included participants from safety analysis set with type 2 diabetes at screening.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 64 | 32
Episodes | 2 | 1

40. Secondary Outcome: Change From Baseline in Pulse
Description: Change in pulse from baseline (week 0) to week 44 is presented. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0), week 44
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment. Overall number of participants analysed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 212 | 98
Beats per minute (bpm) | 4 (10) | 1 (10)

41. Secondary Outcome: Change From Baseline in Amylase: Ratio to Baseline
Description: Change in amylase measured in units/liter (U/L) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0), week 44
Population: as for outcome 40
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 212 | 98
Ratio of amylase | 1.19 (19.4) | 1.08 (20.5)

42. Secondary Outcome: Change From Baseline in Lipase: Ratio to Baseline
Description: Change in lipase measured in units/liter (U/L) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0), week 44
Population: as for outcome 40
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 212 | 98
Ratio of lipase | 1.54 (41.8) | 1.08 (37.8)

43. Secondary Outcome: Change From Baseline in Calcitonin: Ratio to Baseline
Description: Change in calcitonin measured in units/liter (U/L) from baseline (week 0) to week 44 is presented as ratio to baseline. The outcome measure was evaluated based on the data from on-treatment observation period, which was defined as the interval from the date of first trial product administration (week 0) to the date of last trial product administration (week 44) plus a 7 week follow-up period and excluding any off-treatment time intervals.
Time Frame: Baseline (week 0), week 44
Population: as for outcome 40
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of calcitonin
Arm/Group | Semaglutide 2.4 mg | Placebo
Number analyzed (Participants) | 211 | 98
Ratio of calcitonin | 1.04 (37.0) | 0.92 (39.4)

ADVERSE EVENTS:
Time Frame: Week 0 to week 51
Description: All presented AEs are TEAEs, defined as an event with onset during the on-treatment observation period. Results are based on the SAS which included all randomized participants exposed to at least one dose of randomized treatment.
Groups:
- Sema 2.4 mg: Participants initiated at a once weekly dose of 0.25 mg semaglutide s.c. followed a fixed-dose escalation regimen, with dose increasing every 4 weeks (to doses of 0.5, 1.0, 1.7 and 2.4 mg/week), to reach maintenance dose after 16 weeks. Treatment was continued on the maintenance dose of 2.4 mg once-weekly for an additional 28 weeks until week 44 adjunct to a reduced calorie diet and increased physical activity.
Arm/Group | Sema 2.4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/126
Serious Adverse Events (participants affected / at risk) | 14/249 | 8/126
Other Adverse Events (participants affected / at risk) | 180/249 | 57/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sema 2.4 mg (N=249) | Placebo (N=126)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Fascial infection (Infections and infestations) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Thymic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sema 2.4 mg (N=249) | Placebo (N=126)
Abdominal distension (Gastrointestinal disorders) | 25 (34) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 15 (15) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (19) | 3 (3)
COVID-19 (Infections and infestations) | 15 (16) | 5 (5)
Constipation (Gastrointestinal disorders) | 29 (31) | 7 (10)
Decreased appetite (Metabolism and nutrition disorders) | 43 (60) | 5 (8)
Diarrhoea (Gastrointestinal disorders) | 65 (124) | 13 (20)
Dizziness (Nervous system disorders) | 13 (14) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 14 (19) | 0 (0)
Eructation (Gastrointestinal disorders) | 14 (16) | 0 (0)
Nausea (Gastrointestinal disorders) | 60 (78) | 9 (14)
Upper respiratory tract infection (Infections and infestations) | 51 (62) | 26 (34)
Vomiting (Gastrointestinal disorders) | 21 (39) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT04251156/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT04251156/SAP_001.pdf